CLINICAL TRIAL: NCT06427512
Title: Mechanisms Underlying Cardiovascular Consequences Associated With COVID-19 and Long COVID - Characterizing Long COVID Phenotypes Using Physiological and Molecular Studies
Brief Title: Mechanisms Underlying Cardiovascular Consequences Associated With COVID-19 and Long COVID
Status: Withdrawn | Type: Observational
Why Stopped: Funding not available
Sponsor: Columbia University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: AAA-TBA
Record Dates: First submitted 2022-02-01; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: long COVID-19
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID patients: Patients with long COVID-19 and experiencing cardiovascular symptoms at 24 weeks post-acute illness or post-COVID without cardiovascular symptoms by 8 weeks after illness.

SUMMARY:
AIM 1. Characterize cardiovascular phenotypes of long COVID by cardiopulmonary, meta-bolic, and cardiac mechanical/physiological responses to exercise and microvascular vasomotor function.

AIM 2. Identify intercellular signaling between immune cells and cardiac cells associated with microvascular phenotypes of long COVID.

DETAILED DESCRIPTION:
As many as 40-60% of patients who recovered from mild or moderate acute COVID have reported what is now called long COVID - multiple, persistent or recurrent symptoms lasting 6-9 months (or longer) following initial illness.1-4 Fatigue, dyspnea, and chest pain are the most common symptoms. Others include palpitations, lightheadedness, and syncope. All these cardiovascular symptoms can be debilitating, resulting in worse quality of life and morbidity.5, 6 Treatment options are limited.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, < 75 yrs
* History of lab-confirmed COVID
* Symptomatic at >12 wks post-acute COVID (cases)
* Recovered by 8wks post-acute COVID (controls)

Exclusion Criteria:

* Any history of critical illness
* Chronic kidney disease, Stage >4
* Pre-COVID: HFrEF, CABG, arrhythmia; pulmonary hypertension, pulmonary embolus, interstitial lung disease (ILD), O2 dependence; dementia, stroke, autonomic dysfunction; coagulopathy
* Post-COVID: ILD, O2 dependence

Ages: 19 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited primarily from the Prospective COVID-19 ID Persistence Cohort (C-PIC).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Microvascular dysfunction | Up to 2.5 years
  This is to measure the microvascular dysfunction in patients using Cardiac PET.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Tsai, MD, Principal Investigator — Florence Irving Associate Professor of Medicine, Dept of Medicine Cardiology
Locations (1):
- CUIMC, New York, New York, United States

REFERENCES:
- [Background] Blomberg B, Mohn KG, Brokstad KA, Zhou F, Linchausen DW, Hansen BA, Lartey S, Onyango TB, Kuwelker K, Saevik M, Bartsch H, Tondel C, Kittang BR; Bergen COVID-19 Research Group; Cox RJ, Langeland N. Long COVID in a prospective cohort of home-isolated patients. Nat Med. 2021 Sep;27(9):1607-1613. doi: 10.1038/s41591-021-01433-3. Epub 2021 Jun 23. PMID 34163090
- [Background] Nehme M, Braillard O, Alcoba G, Aebischer Perone S, Courvoisier D, Chappuis F, Guessous I; COVICARE TEAM. COVID-19 Symptoms: Longitudinal Evolution and Persistence in Outpatient Settings. Ann Intern Med. 2021 May;174(5):723-725. doi: 10.7326/M20-5926. Epub 2020 Dec 8. No abstract available. PMID 33284676
- [Background] Nehme M, Braillard O, Chappuis F, Courvoisier DS, Guessous I; CoviCare Study Team. Prevalence of Symptoms More Than Seven Months After Diagnosis of Symptomatic COVID-19 in an Outpatient Setting. Ann Intern Med. 2021 Sep;174(9):1252-1260. doi: 10.7326/M21-0878. Epub 2021 Jul 6. PMID 34224254
- [Background] Soriano JB, Murthy S, Marshall JC, Relan P, Diaz JV; WHO Clinical Case Definition Working Group on Post-COVID-19 Condition. A clinical case definition of post-COVID-19 condition by a Delphi consensus. Lancet Infect Dis. 2022 Apr;22(4):e102-e107. doi: 10.1016/S1473-3099(21)00703-9. Epub 2021 Dec 21. PMID 34951953
- [Background] Huang L, Yao Q, Gu X, Wang Q, Ren L, Wang Y, Hu P, Guo L, Liu M, Xu J, Zhang X, Qu Y, Fan Y, Li X, Li C, Yu T, Xia J, Wei M, Chen L, Li Y, Xiao F, Liu D, Wang J, Wang X, Cao B. 1-year outcomes in hospital survivors with COVID-19: a longitudinal cohort study. Lancet. 2021 Aug 28;398(10302):747-758. doi: 10.1016/S0140-6736(21)01755-4. PMID 34454673
- [Background] Sigfrid L, Drake TM, Pauley E, Jesudason EC, Olliaro P, Lim WS, Gillesen A, Berry C, Lowe DJ, McPeake J, Lone N, Munblit D, Cevik M, Casey A, Bannister P, Russell CD, Goodwin L, Ho A, Turtle L, O'Hara ME, Hastie C, Donohue C, Spencer RG, Donegan C, Gummery A, Harrison J, Hardwick HE, Hastie CE, Carson G, Merson L, Baillie JK, Openshaw P, Harrison EM, Docherty AB, Semple MG, Scott JT; ISARIC4C investigators. Long Covid in adults discharged from UK hospitals after Covid-19: A prospective, multicentre cohort study using the ISARIC WHO Clinical Characterisation Protocol. Lancet Reg Health Eur. 2021 Sep;8:100186. doi: 10.1016/j.lanepe.2021.100186. Epub 2021 Aug 6. PMID 34386785